CLINICAL TRIAL: NCT01252966
Title: Cognitive Training for Nicotine Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 812429
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Results first posted 2017-01-02 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Tobacco Use Disorder; Nicotine Addiction
Keywords: Tobacco; Smoking; Cognition; Behavioral Training; Relapse
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Recurrence | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Training (Experimental): Participants in this arm received computerized cognitive training in addition to nicotine patch and smoking cessation counseling.
  Interventions: Behavioral: Cognitive Training
- Control Training (Placebo Comparator): Participants in this arm received computerized control training in addition to nicotine patch and smoking cessation counseling
  Interventions: Behavioral: Control training

INTERVENTIONS:
Behavioral: Cognitive Training — The computerized cognitive training intervention is a 12-week standardized course of internet-based computerized cognitive exercises designed to enhance executive cognitive function.
  Arms: Cognitive Training
Behavioral: Control training — The computerized control training intervention is a 12-week standardized course of internet-based deep breathing exercises which does not contain the cognitive exercises designed to enhance executive cognitive function.
  Arms: Control Training

SUMMARY:
This randomized clinical trial tested the effects of a computerized (web-based) cognitive training intervention on smoking cessation.

All participants received 8 weeks of standard nicotine patch therapy, smoking cessation counseling, and were randomized to 1 of 2 different training programs: cognitive training vs. control training.

ELIGIBILITY:
Inclusion:

1. Healthy male and female treatment-seeking smokers who are between 18 and 65 years of age and self-report smoking at least 5 cigarettes (menthol and/or non-menthol) per day for at least the last 6 months
2. Plan to live in the area for at least the next 8 months
3. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form
4. Able to communicate fluently in English (speaking, writing, and reading)
5. Have uninterrupted access to a home computer with sound capabilities, keyboard, mouse, and active Internet connection
6. Provide a Carbon Monoxide (CO) breath test reading greater than or equal to 8 parts per million (ppm) at Intake Visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2011-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caryn Lerman, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Interdiscplinary Research on Nicotine Addiction, University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Kable JW, Caulfield MK, Falcone M, McConnell M, Bernardo L, Parthasarathi T, Cooper N, Ashare R, Audrain-McGovern J, Hornik R, Diefenbach P, Lee FJ, Lerman C. No Effect of Commercial Cognitive Training on Brain Activity, Choice Behavior, or Cognitive Performance. J Neurosci. 2017 Aug 2;37(31):7390-7402. doi: 10.1523/JNEUROSCI.2832-16.2017. Epub 2017 Jul 10. PMID 28694338

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this clinical trial began in March 2011. Study accrual was completed in September 2015, with a final sample of N=213 in the intention-to-treat (ITT) analysis.
Pre-assignment Details: Five hundred and fifty-seven participants provided consent and 213 were randomized. Reasons for exclusion from randomization included no home computer or internet access and failure to meet final eligibility criteria at the Intake Visit.
Groups:
- Cognitive Training: The Cognitive Training intervention is a 12-week standardized course of internet-based computerized cognitive exercises designed to enhance executive cognitive function. Participants also receive nicotine patch and smoking cessation counseling.
- Control Training: The Control Training intervention is a 12-week standardized course of internet-based deep breathing exercises which does not contain the cognitive exercises designed to enhance executive cognitive function. Participants also receive nicotine patch and smoking cessation counseling.
Period: Overall Study
Arm/Group | Cognitive Training | Control Training
Started | 108 | 105
Completed | 85 | 92
Not Completed | 23 | 13
Not completed — Lost to Follow-up | 16 | 10
Not completed — Withdrawal by Subject | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Training | Control Training | Total
Number analyzed (Participants) | 108 | 105 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.18 (12.62) | 43.39 (12.38) | 43.28 (12.48)
Gender [Count of Participants; unit: Participants]
  Female | 53 | 54 | 107
  Male | 55 | 51 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 107 | 100 | 207
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 38 | 42 | 80
  White | 61 | 54 | 115
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 108 | 105 | 213
Cigarettes Per Day [Mean (Standard Deviation); unit: cigarettes smoked per day] | 16.42 (6.14) | 15.73 (5.23) | 16.08 (5.70)
Fagerström Test for Nicotine Dependence Score [Mean (Standard Deviation); unit: units on a scale] — The Fagerström Test for Nicotine Dependence (FTND) will be administered; this is a 6-item measure of nicotine dependence which has good internal consistency and high test-retest reliability (r=.88). Scores may range from 0 to 9, with higher scores indicating greater nicotine dependence.
  units on a scale | 4.82 (2.11) | 4.65 (1.74) | 4.74 (1.94)

OUTCOME MEASURES:

1. Primary Outcome: Point-prevalence Abstinence at End of Treatment
Description: Daily smoking, from the Target Quit Date to End of Treatment (EOT), was assessed by a validated timeline follow-back measure. Based on guidelines for smoking cessation trials, the primary outcome was 7-day point prevalence abstinence at EOT, and abstinence was defined as no self-reported smoking (even a puff) for at least 7 days, with in-person verification by carbon monoxide breath levels (CO <8ppm). Following standard convention, participants who withdrew or were lost to follow-up were considered smokers.
Time Frame: End of treatment (Week 12)
Measure: Number; unit: Percentage of participants
Arm/Group | Cognitive Training | Control Training
Number analyzed (Participants) | 108 | 105
Percentage of participants | 38 | 43
Statistical Analysis 1: Comparison: Cognitive Training vs Control Training; Longitudinal logistic regression with fitted generalized estimating equations (GEE) was used to estimate an overall treatment effect odds ratio including both the EOT and 6-month time points and relevant covariates (e.g., baseline smoking rate, age, Shipley IQ score). The study (n=213) had 80% power to detect small to medium effects on quit rates (corresponding to Cohen's one-sample d=0.38); Test type: Superiority or Other; p = 0.14, Regression, Logistic; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.42 to 1.13]

2. Secondary Outcome: Point-prevalence Abstinence at 6-month Follow-up
Description: Daily smoking from the Target Quit Date to 6 month follow-up was assessed by a validated timeline follow-back measure. Based on guidelines for smoking cessation trials, the secondary outcome was 7-day point prevalence abstinence at the 6 month follow-up, and abstinence was defined as no self-reported smoking (even a puff) for at least 7 days, with in-person verification by carbon monoxide breath levels (CO <8ppm). Following standard convention, participants who withdrew or were lost to follow-up were considered smokers.
Time Frame: 6 month follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | Cognitive Training | Control Training
Number analyzed (Participants) | 108 | 105
Percentage of participants | 15 | 25

3. Secondary Outcome: Cognitive Performance (Working Memory)
Description: Change in performance on the Digit Span Forward task (working memory) between Baseline and End of Treatment (Week 12). In this task, participants are presented with a series of digits on the computer screen at one second intervals. Participants are then required to enter the digits in order. The number of digits in each series ranges from 3 to 7, and the maximum recall span is the length of the largest series entered correctly. The outcome measure is the change score (calculated by subtracting the Baseline score from the end of treatment score). Change scores can range from -4 to 4. Negative numbers indicate worse performance at EOT; positive numbers indicate better performance at EOT; and 0 indicates no change.
Time Frame: Baseline and Week 12 (EOT)
Population: Participants with performance >3SD from the mean at baseline were excluded as outliers.
Measure: Mean (Standard Deviation); unit: Change in maximum recall span
Arm/Group | Cognitive Training | Control Training
Number analyzed (Participants) | 82 | 92
Change in maximum recall span | 0.22 (1.2) | 0.03 (1.1)
Statistical Analysis 1: Comparison: Cognitive Training vs Control Training; Multiple regression models were used to estimate effects of treatment on change in cognitive performance. Age, Shipley IQ score, number of cigarettes smoked per day at baseline, and EOT smoking status were included as covariates; Test type: Superiority or Other; p = 0.30, Regression, Linear

4. Secondary Outcome: Cognitive Performance (Response Inhibition)
Description: Change in performance on the Go/No-Go Task (response inhibition) between Baseline and End of Treatment (Week 12). In this task, participants are presented with a series of stimuli (the word "PRESS" in either green or red). Participants are instructed to respond by pressing the spacebar when the stimulus is green, and to withhold a response when the stimulus is red. The outcome is the change in number of commission errors (failure to withhold a response to a red stimulus) from EOT minus baseline. The potential range for the change score is -42 to 42. Negative numbers indicate a decrease in the number of commission errors (improved performance) from baseline to EOT; positive numbers indicate an increase in commission errors (worse performance); 0 indicates no change.
Time Frame: Baseline and Week 12 (EOT)
Population: Participants with performance >3SD from the mean at baseline were excluded as outliers.
Measure: Mean (Standard Deviation); unit: Change in number of commission errors
Arm/Group | Cognitive Training | Control Training
Number analyzed (Participants) | 82 | 92
Change in number of commission errors | -0.84 (2.5) | -0.49 (2.5)
Statistical Analysis 1: Comparison: Cognitive Training vs Control Training; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.30, Regression, Linear

5. Secondary Outcome: Cognitive Performance (Attention)
Description: Change in performance on the Continuous Performance Task (attention) between Baseline and End of Treatment (Week 12). In this task, participants are presented with a series of letters at 2.5s intervals and are instructed to respond by pressing the space bar if the same letter appears twice in a row. The outcome is the change in the number of commission errors (the number of times the participant responded to a non-target at EOT minus baseline). There are a total of 125 trials, with 20 target trials (response required) and 85 non-target trials (no response required); therefore the possible range for the change score is -85 to 85. Negative numbers indicate a decrease in commission errors (better performance at EOT compared to baseline); positive numbers indicate an increase in commission errors (worse performance at EOT compared to baseline); and 0 indicates no change.
Time Frame: Baseline and Week 12 (EOT)
Population: Participants with performance >3SD from the mean at Baseline were excluded as outliers.
Measure: Mean (Standard Deviation); unit: Change in number of commission errors
Arm/Group | Cognitive Training | Control Training
Number analyzed (Participants) | 82 | 92
Change in number of commission errors | -0.27 (1.3) | 0.54 (1.6)
Statistical Analysis 1: Comparison: Cognitive Training vs Control Training; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.033, Regression, Linear — Results would not survive correction for multiple hypothesis testing

ADVERSE EVENTS:
Time Frame: AE and SAE data were collected from enrollment through follow up (~31 weeks).
Description: Participants (PPTs) completed an anticipated side effects questionnaire (transdermal nicotine) at Pre-Quit (baseline measure) and at every subsequent in-person visit during the treatment period (systematic assessment). AE and SAE information was collected via spontaneous report from enrollment through follow up as a non-systematic assessment (n=213).
Arm/Group | Cognitive Training | Control Training
Serious Adverse Events (participants affected / at risk) | 6/108 | 3/105
Other Adverse Events (participants affected / at risk) | 42/108 | 54/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Training (N=108) | Control Training (N=105)
Squamous Cell Carcinoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Squamous cell carcinoma was treated by surgical excision. The procedure was successful in removal of the Squamous Cell Carcinoma.
Infection (Infections and infestations) | 1 (1) | 0 (0) — Ppt admitted to the hospital due to a severe infection at the site of a root canal.
Pancreatitis (General disorders) | 1 (1) | 0 (0)
Emergency Procedure (Surgical and medical procedures) | 1 (1) | 0 (0) — PPT complaining of chest/neck pain. PPT was dx with CAD and underwent an emergency procedure to implant 2 stents.
Bowel Blockage (Gastrointestinal disorders) | 1 (1) | 0 (0) — Ppt was admitted to the hospital for treatment.
Collapsed Lung (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Breast Cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1) — PPT was dx. with Stage 4 Breast Cancer and underwent radiation tx.
Surgery (Gastric Bypass) (Surgical and medical procedures) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Training (N=108) | Control Training (N=105)
Headache (Nervous system disorders) | 10 (11) | 12 (12)
Nausea (Gastrointestinal disorders) | 6 (6) | 6 (6)
Insomnia (Psychiatric disorders) | 22 (35) | 37 (59)
Skin Irritation (Skin and subcutaneous tissue disorders) | 8 (11) | 13 (13)
Sweating (Skin and subcutaneous tissue disorders) | 5 (9) | 7 (7)
Disturbing Dreams (Psychiatric disorders) | 10 (10) | 12 (13)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes